CLINICAL TRIAL: NCT01649284
Title: LUX-Lung EAP US; An Open Label Expanded Access Program of Afatinib (BIBW 2992) for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring EGFR Mutation(s)
Brief Title: Afatinib Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.45
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

INTERVENTIONS:
Drug: afatinib — 40, 30, and 20 mg film-coated tablets

SUMMARY:
This is an open-label, multi-center, single-arm trial, designed to provide early access to afatinib and to provide additional information on the safety and efficacy of afatinib in advanced NSCLC patients who harbor an EGFR mutation.

ELIGIBILITY:
Inclusion criteria:

Patients with:

1. locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC)
2. Epidermal Growth Factor Receptor (EGFR) mutation-positive result per the institution's testing methodology.
3. male or female patients age >=18 years
4. Adequate organ function, defined as all of the following:

   1. Left Ventricular Ejection Fraction (LVEF) >50% or within institution normal values
   2. Absolute Neutrophil Count (ANC) > 1500/mm3.
   3. Platelet count >75,000/mm3
   4. Serum creatinine < 1.5 times of the upper limit of normal
   5. Total Bilirubin < 1.5 times upper limit of (institutional) normal.
   6. Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) < three times the upper limit of (institutional) normal (ULN).
5. ECOG score between 0 - 2
6. written informed consent by patient or guardian prior to admission into the trial that is consistent with International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP) guidelines and local law.

Exclusion criteria:

Patients who or with:

1. hormonal anti-cancer treatment within 2 weeks prior to start of trial treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted)
2. Radiotherapy within 14 days prior to drug administration, except as follows:

   1. Palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
   2. Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
3. major surgery within 4 weeks before starting trial treatment or scheduled for surgery during the projected course of the trial
4. known hypersensitivity to afatinib or any of its excipients
5. history or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia as determined by the treating physician. Myocardial infarction within 6 months prior to starting trial treatment.
6. are Women of Child-Bearing Potential (WOCBP) and men who are able to father a child, unwilling to be abstinent or use adequate contraception prior to trial entry, for the duration of trial participation and for at least 2 weeks after treatment has ended.
7. childbearing potential who are: a) are nursing or b) are pregnant or c) are not using an acceptable method of birth control, or do not plan to continue using this method throughout the trial and/or do not agree to submit to pregnancy testing required by this protocol
8. any history of or concomitant condition that, in the opinion of the treating physician, would compromise the patient's ability to comply with the trial or interfere with the evaluation of safety for the trial drug
9. previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
10. requiring treatment with any of the prohibited concomitant medications listed in Section 4.2.2 of the protocol that can not be stopped for the duration of trial participation
11. known pre-existing interstitial lung disease
12. presence of poorly controlled gastrointestinal disorders that could affect the absorption of the trial drug based on treating physician assessment.
13. active hepatitis B infection, active Hepatitis C (HEP C) infection and/or known Human Immunodeficiency Virus (HIV) carrier.
14. meningeal carcinomatosis
15. symptomatic brain metastases (patients with asymptomatic brain metastases, who were previously treated, are eligible provided they have had Stable Disease (SD) for at least 4 weeks on stable doses of medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (66):
- United States (66):
  - 1200.45.004 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1200.45.116 Boehringer Ingelheim Investigational Site, Goodyear, Arizona
  - 1200.45.057 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1200.45.078 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1200.45.114 Boehringer Ingelheim Investigational Site, Burbank, California
  - 1200.45.123 Boehringer Ingelheim Investigational Site, Glendale, California
  - 1200.45.115 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1200.45.117 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1200.45.102 Boehringer Ingelheim Investigational Site, Monterey, California
  - 1200.45.091 Boehringer Ingelheim Investigational Site, Pleasant Hill, California
  - 1200.45.098 Boehringer Ingelheim Investigational Site, Pleasant Hill, California
  - 1200.45.006 Boehringer Ingelheim Investigational Site, Ranco Cucamonga, California
  - 1200.45.003 Boehringer Ingelheim Investigational Site, Southington, Connecticut
  - 1200.45.007 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1200.45.026 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1200.45.097 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1200.45.017 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1200.45.058 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1200.45.016 Boehringer Ingelheim Investigational Site, Lakeland, Florida
  - 1200.45.103 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 1200.45.037 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1200.45.056 Boehringer Ingelheim Investigational Site, Port Saint Lucie, Florida
  - 1200.45.119 Boehringer Ingelheim Investigational Site, Titusville, Florida
  - 1200.45.095 Boehringer Ingelheim Investigational Site, Alpharetta, Georgia
  - 1200.45.029 Boehringer Ingelheim Investigational Site, Athens, Georgia
  - 1200.45.042 Boehringer Ingelheim Investigational Site, Macon, Georgia
  - 1200.45.121 Boehringer Ingelheim Investigational Site, Valdosta, Georgia
  - 1200.45.024 Boehringer Ingelheim Investigational Site, Decatur, Illinois
  - 1200.45.009 Boehringer Ingelheim Investigational Site, Evanston, Illinois
  - 1200.45.099 Boehringer Ingelheim Investigational Site, Peoria, Illinois
  - 1200.45.040 Boehringer Ingelheim Investigational Site, Waterloo, Iowa
  - 1200.45.041 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1200.45.083 Boehringer Ingelheim Investigational Site, Marrero, Louisiana
  - 1200.45.087 Boehringer Ingelheim Investigational Site, Metairie, Louisiana
  - 1200.45.019 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1200.45.039 Boehringer Ingelheim Investigational Site, Rockville, Maryland
  - 1200.45.053 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1200.45.046 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1200.45.100 Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - 1200.45.067 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1200.45.071 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 1200.45.021 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1200.45.066 Boehringer Ingelheim Investigational Site, Freehold, New Jersey
  - 1200.45.105 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1200.45.080 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1200.45.068 Boehringer Ingelheim Investigational Site, Fresh Meadows, New York
  - 1200.45.051 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.45.092 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.45.001 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1200.45.086 Boehringer Ingelheim Investigational Site, Bismarck, North Dakota
  - 1200.45.048 Boehringer Ingelheim Investigational Site, Minot, North Dakota
  - 1200.45.090 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1200.45.005 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1200.45.089 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1200.45.094 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1200.45.020 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1200.45.096 Boehringer Ingelheim Investigational Site, Johnstown, Pennsylvania
  - 1200.45.060 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1200.45.085 Boehringer Ingelheim Investigational Site, Pottstown, Pennsylvania
  - 1200.45.120 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 1200.45.049 Boehringer Ingelheim Investigational Site, Cookeville, Tennessee
  - 1200.45.113 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 1200.45.045 Boehringer Ingelheim Investigational Site, Fairfax, Virginia
  - 1200.45.076 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 1200.45.093 Boehringer Ingelheim Investigational Site, Charleston, West Virginia
  - 1200.45.125 Boehringer Ingelheim Investigational Site, Wausau, Wisconsin

REFERENCES:
- [Derived] Kim ES, Halmos B, Kohut IF, Patel T, Rostorfer RD, Spira AI, Cseh A, McKay J, Wallenstein G, Mileham KF. Efficacy and Safety Results of the Afatinib Expanded Access Program. Oncol Ther. 2017;5(1):103-110. doi: 10.1007/s40487-017-0043-5. Epub 2017 Apr 10. PMID 28680960